CLINICAL TRIAL: NCT02332486
Title: Based on Metabonomics Dryness Pathogen Type of Oral Lichen Planus of Dynamic
Brief Title: Based on Metabonomics Dryness Pathogen Type of OLP: a Dynamic Study
Acronym: OLP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yang Xuyan, Deputy director of First Affiliated Hospital of Heilongjiang University of Chinese Medicine Department of Stomatology, Heilongjiang University of Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OLP-Metabonomics-2014; 81403441 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2014-12-30; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Jiawei qingxuan jiangya decoction

ARMS (2):
- Intervene (Active Comparator): For Qingxuan Decoction there are a bag of Chinese honeylocust spine，Glehnia littoralis and Smilax china L,and two bags of Silktree albizia bark, Kadsura interior,Cortex dictamni, Lilium brownii var, Silkworm larva,Forsythia suspensa and Rhizoma polygonati preparata, and three bags of viridulumArisaema erubescens and Poria cocos Wolf. All drugs are made by Jiangyin Tianjiang company in China. Qingxuan Decoction is given two times after breakfast and dinner in 56 days.
  Interventions: Drug: Qingxuan Decoction
- Blank (No Intervention): There is no intervention for people in the blank group.

INTERVENTIONS:
Drug: Qingxuan Decoction — In Qingxuan Decoction, there are a bag of Chinese honeylocust spine，Glehnia littoralis and Smilax china L,and two bags of Silktree albizia bark, Kadsura interior,Cortex dictamni, Lilium brownii var, Silkworm larva,Forsythia suspensa and Rhizoma polygonati preparata, and three bags of viridulumArisaema erubescens and Poria cocos Wolf. All drugs are made by Jiangyin Tianjiang company in China.
  Arms: Intervene

SUMMARY:
Due to the change of life style, the incidence of oral cavity mucous membrane disease increased.In this study，been done a large number of pre-clinical practice and some experimental studies， based on the application of metabolomics technology to ultra-high liquid-mass spectrometry metabolomics analyzer as the core means， The metabolism of pattern recognition and combination of modern analytical techniques to measure blood and urine of patients with OLP-specific clearance of endogenous metabolites，and after the intervention of moss drink endogenous metabolites in the body as a whole group of. At the same time， the use of flow cytometry,，ELISA， immunohistochemistry and other modern technology, research OLP patients using clean moss drink before and after treatment of local lesions and peripheral blood CD4 +，CD8 + lymphocytes，Th1 cytokines (IFN-γ， TNF-α)， Th2 cytokines (IL-4，10) the dynamic changes. From metabolomics， cellular immunology， inflammation mechanism perspective of local OLP lesions， peripheral blood and changes in endogenous metabolites in the process,，in-depth study of traditional Chinese medicine to drink clean moss multi-component multi-target treatment of this disease mechanism， is widely used in traditional Chinese medicine treatment of OLP provide a theoretical basis for the promotion of Chinese medicine Qingxian Yin in the oral mucosal disease in the application， effectively solve clinical practice problems.

ELIGIBILITY:
Inclusion Criteria:

* All patients with OLP .
* TCM syndrome of OLP patients included is dryness pathogen type.
* In the lesions of oral mucosa there are phanerous pearly white keratinization stripes, or patches, or phanerous erosion with the mucous membrane hyperemia.
* OLP patients may accompany oral coarse discomfort or pain, red tongue, yellow dry or dry fur, dry mouth, bitter taste.

Exclusion Criteria:

* Patients with other established oral mucosal disease;
* Patients accompanied by serious systemic diseases, eg damaged liver or kidney functions; Or other allergic diseases, eg rheumatic disease or cancer.
* Patients using the antibiotic in the last one month or immunologic agents in the last three months.
* Lichenoid reaction caused by drugs or the filling with silver and amalgam.
* Patients with smoking or alcoholism in the last three months.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
visualanalogue scale | every week of eight weeks

SECONDARY OUTCOMES:
Cytokines | every week of eight weeks
  IFN-γ, TNF-α, IL-4 and IL-10 of the blood cells of CD4+/CD8+ and Th1/Th2 will be tested by flow cytometry or ELISA.
Cytokines | rvery week of eight weeks
  IFN-γ, TNF-α, IL-4 and IL-10 of the lesion tissue cells of CD4+/CD8+ and Th1/Th2 will be tested by immunohistochemistry
Biomarker | every week of eight weeks
  Metabolites profiles of individual in the intervention group will be analysed by PCA、OPLS-DA or UPLC-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xu Yan, Doctor, Principal Investigator — University of Chinese Medicine Department of Stomatology, Heilongjiang University of Chinese Medicine.

REFERENCES:
- [Result] Scully C, Carrozzo M. Oral mucosal disease: Lichen planus. Br J Oral Maxillofac Surg. 2008 Jan;46(1):15-21. doi: 10.1016/j.bjoms.2007.07.199. Epub 2007 Sep 5. PMID 17822813
- [Result] Holmstrup P, Thorn JJ, Rindum J, Pindborg JJ. Malignant development of lichen planus-affected oral mucosa. J Oral Pathol. 1988 May;17(5):219-25. doi: 10.1111/j.1600-0714.1988.tb01528.x. PMID 3144585
- [Result] Gandolfo S, Richiardi L, Carrozzo M, Broccoletti R, Carbone M, Pagano M, Vestita C, Rosso S, Merletti F. Risk of oral squamous cell carcinoma in 402 patients with oral lichen planus: a follow-up study in an Italian population. Oral Oncol. 2004 Jan;40(1):77-83. doi: 10.1016/s1368-8375(03)00139-8. PMID 14662419
- [Result] Chaiyarit P, Ma N, Hiraku Y, Pinlaor S, Yongvanit P, Jintakanon D, Murata M, Oikawa S, Kawanishi S. Nitrative and oxidative DNA damage in oral lichen planus in relation to human oral carcinogenesis. Cancer Sci. 2005 Sep;96(9):553-9. doi: 10.1111/j.1349-7006.2005.00096.x. PMID 16128740
- [Result] Mosmann TR, Cherwinski H, Bond MW, Giedlin MA, Coffman RL. Two types of murine helper T cell clone. I. Definition according to profiles of lymphokine activities and secreted proteins. 1986. J Immunol. 2005 Jul 1;175(1):5-14. No abstract available. PMID 15972624
- [Result] Lee YC. Synergistic effect of various regulatory factors in TH1/TH2 balance; immunotherapeutic approaches in asthma. Int J Biomed Sci. 2008 Mar;4(1):8-13. PMID 23675060
- [Result] Krouwels FH, van der Heijden JF, Lutter R, van Neerven RJ, Jansen HM, Out TA. Glucocorticosteroids affect functions of airway- and blood-derived human T-cell clones, favoring the Th1 profile through two mechanisms. Am J Respir Cell Mol Biol. 1996 Apr;14(4):388-97. doi: 10.1165/ajrcmb.14.4.8600944.
- [Result] Agarwal SK, Marshall GD Jr. Dexamethasone promotes type 2 cytokine production primarily through inhibition of type 1 cytokines. J Interferon Cytokine Res. 2001 Mar;21(3):147-55. doi: 10.1089/107999001750133159. PMID 11331037
- [Result] van der Meij EH, van der Waal I. Lack of clinicopathologic correlation in the diagnosis of oral lichen planus based on the presently available diagnostic criteria and suggestions for modifications. J Oral Pathol Med. 2003 Oct;32(9):507-12. doi: 10.1034/j.1600-0714.2003.00125.x. PMID 12969224
- [Result] Mendoza L. A network model for the control of the differentiation process in Th cells. Biosystems. 2006 May;84(2):101-14. doi: 10.1016/j.biosystems.2005.10.004. Epub 2005 Dec 28. PMID 16386358